CLINICAL TRIAL: NCT01958125
Title: A Randomized, Multicentre, Double-blind, Parallel, Sham-controlled Study of GammaCore®, a Non-invasive Neurostimulator Device for the Acute Relief of Episodic and Chronic Cluster Headache.
Brief Title: A Randomized Multicentre Study for the Acute Relief of Episodic and Chronic Cluster Headache.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GC-003
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cluster Headache
Keywords: vagus nerve stimulation; vagal nerve stimulation; nVNS; VNS; cluster headache; non invasive; gammacore
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gammacore (Active Comparator): gammacore active device to be used noninvasively to the vagal nerve in the neck.
  Interventions: Device: gammaCore
- inactive gammacore (Placebo Comparator): same as the active treatment, but without the therapy treatment provided
  Interventions: Device: gammaCore

INTERVENTIONS:
Device: gammaCore — Vagal stimulation

SUMMARY:
The study will look at a non-invasive treatment for people suffering with chronic and episodic headaches. Study subjects will be randomized to an active treatment or an in-active treatment for 2 weeks. After the 2 weeks all subjects will continue to treat with an active treatment for an additional 2 weeks.

DETAILED DESCRIPTION:
The study is a prospective double blind, randomized, sham-controlled, multi-center investigation designed for comparison of two parallel groups, GammaCore® (active treatment) and a sham, (in-active) treatment. The study period begins with a 1-week run-in period, followed by a 2 week comparative period when the subjects are randomized (1:1) to either active treatment or sham (in-active) treatment. The comparative period will be followed by an open label 2 week period, where the subjects in the sham treatment group will switch in treatment assignment and receive an active treatment and the active group will continue to receive an active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years or older
* Has been diagnosed with episodic or chronic cluster headache in accordance with the ICHD-2 Classification criteria (2ndEd)
* Is capable of completing the 5-point pain scale, disability scale and other self-assessments
* Agrees to refrain from starting new medication aimed to control the cluster headache for the duration of the run-in and randomized phase
* Is able to provide written Informed Consent

Exclusion Criteria:1.

* Episodic cluster headache sufferers who are not in a cluster headache bout at the time of screening and enrollment
* 2. Need to commence treatment with oral or injectable steroids for eventual concomitant medical conditions
* 3. Has a lesion (including lymphadenopathy), dysaesthesia, previous surgery or abnormal anatomy at the GammaCore® treatment site
* 4. Is currently taking medication for indications other than CH that in the opinion of the clinician may interfere with the study
* 5. Has a history of any cranial aneurysm, intracranial haemorrhage, brain tumours or significant head trauma
* 6. Diagnosed or suspected secondary headache
* 7. Has other significant pain problem that might confound the study assessments in the opinion of the investigator
* 8. Has known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (e.g. bruits or history of transient ischemic attack (TIA) or cerebral vascular accident CVA), congestive heart failure (CHF), known severe coronary artery disease or recent (5 years) myocardial infarction
* 9. Has an abnormal baseline ECG (e.g. second and third degree heart block, atrial fibrillation, atrial flutter, recent history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction)
* 10. Has had a previous, cervical vagotomy
* 11. Has uncontrolled high blood pressure
* 12. Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant
* 13. Has a history of carotid endarterectomy or vascular neck surgery
* 14. Has been implanted with metal cervical spine hardware or has a metallic implant near the GammaCore stimulation site
* 15. Has a recent (12 months) or repeated history of syncope
* 16. Has a recent (12 months) or repeated history of seizure
* 17. Has a known history or suspicion of substance abuse or addiction, or overuse of acute headache medication
* 18. Has psychiatric or cognitive disorder and/or behavioural problems which in the opinion of the clinician may interfere with the study
* 19. Is pregnant, nursing, thinking of becoming pregnant in the next 6 weeks 20. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days
* 21. Is a relative of or an employee of the investigator or the clinical study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Goadsbury, Prof., Principal Investigator — Royal Free Hospital, Dept for Neurology and Clinical Neurosciences
Locations (9):
- Glostrup Hospital, Danish Headache Centre, Glostrup Municipality, Denmark
- Germany (3):
  - Westdeutches Kopfschmerzzentrum, Essen
  - Kopfschmerzklinik Königstein, Königstein im Taunus
  - Klinikum Grosshadern, University of Munich, Munich
- Leiden University Medical Center, Neurology Department, K5-Q-104, Leiden, Netherlands
- United Kingdom (4):
  - Hull Royal Infirmary, Neurology Department, Hull, East Yorkshire
  - Royal Free, Dept for Neurology and Clinical Neurosciences, London, Greater London
  - The Southern Hospital, Neurology Department, Glasgow, Lanarkshire
  - The Walton Center, Neurology Department, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: No
The study is publlished and no other IPD data will be shared.

REFERENCES:
- [Derived] de Coo IF, Marin JC, Silberstein SD, Friedman DI, Gaul C, McClure CK, Tyagi A, Liebler E, Tepper SJ, Ferrari MD, Goadsby PJ. Differential efficacy of non-invasive vagus nerve stimulation for the acute treatment of episodic and chronic cluster headache: A meta-analysis. Cephalalgia. 2019 Jul;39(8):967-977. doi: 10.1177/0333102419856607. Epub 2019 Jun 10. PMID 31246132
- See also: Non-invasive vagus nerve stimulation for the acute treatment of episodic and chronic cluster headache: A randomized, double-blind, sham-controlled ACT2 study. — http://www.ncbi.nlm.nih.gov/pubmed/29231763

RESULTS

PARTICIPANT FLOW:
Groups:
- gammaCore: Active Comparator: gammacore gammacore active device to be used noninvasively to the vagal nerve in the neck
- Sham Device: Placebo Comparator: inactive gammacore same as the active treatment, but without the therapy treatment provided
Period: Overall Study
Arm/Group | gammaCore | Sham Device
Started | 50 | 52
Completed | 48 | 44
Not Completed | 2 | 8
Not completed — Missing diary data | 2 | 6
Not completed — No headache attacks | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | gammaCore | Sham Device | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 52 | 101
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (10.60) | 46.9 (10.63) | 45.4 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 35 | 38 | 73
Region of Enrollment [Number; unit: participants]
  Netherlands | 16 | 14 | 30
  Denmark | 2 | 2 | 4
  United Kingdom | 25 | 27 | 52
  Germany | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Headache Pain Free Attack Rates at 15 Minutes Following the Treatment
Description: Headache pain was collected at the beginning of the attack (all treated attacks) and 15 minutes post treatment pain free attacks.
  Data was collected in the patient diary.
Time Frame: 2 weeks
Population: ITT-Intention To Treat population
Measure: Number; unit: Number of attacks
Arm/Group | gammaCore | Sham Device
Number analyzed (Participants) | 48 | 44
Number of attacks
  Number of treated attacks | 495 | 400
  Number of treated attack pain free at 15 minutes | 67 | 46

2. Secondary Outcome: Change in Disability From Baseline (Randomization) to 2 Weeks After Baseline
Description: Mean difference of scores on a 5 step disability scale. Disability was measured at baseline and after the randomization phase (2 weeks later). Lowest score is 1 and is better than the higher score at 5 that is the worst. An increase, higher scores, means worsening.
  1. minor
  2. minor/moderate
  3. moderate
  4. moderate/severe
  5. severe
Time Frame: 2 weeks
Population: Safety population, three patients in the Sham device group have no data
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | gammaCore | Sham Device
Number analyzed (Participants) | 50 | 49
units on a scale
  Disability score at baseline | 3.9 (0.2) | 3.7 (0.2)
  Disability score at 2 weeks | 3.3 (0.2) | 3.2 (0.2)

3. Secondary Outcome: Mean Change of Questionnaire EQ-5D-3L (Euroqol- 5D-3L) From Baseline to After 2 Weeks Treatment
Description: EQ-5D-3L descriptive system comprises 5 dimensions: mobility, self-care, activity, pain and anxiety. Each dimension has 3 levels: 1 = no problems, 2 = moderate problems, 3=extreme problems. Subjects indicate health state by ticking choosing appropriate statement in each dimension and a VAS scale (Overall health) from 0-100 mm where higher score is better (100) than lower score (0).
  Patients completed the EQ-5D-3L at baseline (the start of the randomized period and at 2 weeks).
Time Frame: 2 weeks
Population: Safety population, three patients in the Sham group had no data for EQ-5D-3L
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | gammaCore | Sham Device
Number analyzed (Participants) | 50 | 49
units on a scale
  Mobility at baseline | 1.2 (0.1) | 1.2 (0.1)
  Mobility after 2 weeks | 1.3 (0.1) | 1.1 (0.1)
  Selfcare at baseline | 1.1 (0) | 1.1 (0)
  Selfcare after 2 weeks | 1.1 (0) | 1.1 (0)
  Activity baseline | 1.7 (0.1) | 1.6 (0.1)
  Activity after 2 weeks | 1.6 (0.1) | 1.6 (0.1)
  Pain at baseline | 2.1 (0.1) | 1.9 (0.1)
  Pain after 2 weeks | 1.7 (0.1) | 1.8 (0.1)
  Anxiety at baseline | 1.5 (0.1) | 1.6 (0.1)
  Anxiety after 2 weeks | 1.3 (0.1) | 1.5 (0.1)
  VAS scale at baseline | 58.9 (2.5) | 63.7 (2.1)
  VAS scale after 2 weeks | 61.4 (2.5) | 66.5 (2.1)

4. Secondary Outcome: Patients Who Used Any Type of Rescue Medication
Description: Following treatment at 15 minutes, patients recorded use of any rescue medication(s) in the diary'
Time Frame: 2 weeks
Population: ITT-Intention To Treat population
Measure: Number; unit: participants
Arm/Group | gammaCore | Sham Device
Number analyzed (Participants) | 48 | 44
participants | 40 | 42

5. Secondary Outcome: Comparison of the Headache Pain Free Attack Rates at 30 Minutes Following the Treatment
Description: The headache pain was collected at the beginning of the attack and 30 minutes post treatment in the patient diary.
  The number of pain free (no pain) attacks are compared to all attacks treated
Time Frame: 2 weeks
Population: ITT-Intention To Treat population
Measure: Number; unit: Number of attacks
Arm/Group | gammaCore | Sham Device
Number analyzed (Participants) | 48 | 44
Number of attacks
  Number of attacks treated | 495 | 400
  Number of attacks treated and pain free at 30 min. | 101 | 81

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: diaries and open questions
Arm/Group | gammaCore | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/52
Other Adverse Events (participants affected / at risk) | 20/50 | 14/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gammaCore (N=50) | Sham Device (N=52)
Left lower pain abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0) — Abdominal pain
Depressed and anxious (Psychiatric disorders) | 0 (0) | 1 (2) — Patient experienced more anxiety and depression after starting treatment
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gammaCore (N=50) | Sham Device (N=52)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain lowe (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Application site irritation (General disorders) | 2 (2) | 0 (0)
Application site paraesthesia (General disorders) | 2 (2) | 1 (1)
Application site vesicles (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myokymia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Typical aura without headache (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Piloerection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin sensitisation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less